CLINICAL TRIAL: NCT02227927
Title: Treatment Use of Domperidone for Gastroparesis
Status: No longer available | Type: Expanded Access
Sponsor: Scott Gabbard, MD (Other)
Responsible Party: Sponsor-Investigator, Scott Gabbard, MD, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: CCF-Domperidone; CCF-Domperidone (Other: Cleveland Clinic)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Gastroparesis
Keywords: Gastroesophageal Reflux Disease; GERD; Gastroparesis; Domperidone
MeSH Terms: conditions — Gastroesophageal Reflux; Gastroparesis | interventions — Domperidone

INTERVENTIONS:
Drug: Domperidone — 10-30mg oral dose, four times daily.

SUMMARY:
Domperidone is a drug that may be of benefit to individuals with gastroesophageal reflux disease (GERD), with upper GI symptoms, gastroparesis, and chronic constipation.

This is a long-term treatment program for prescription of this drug to all patients who, in the investigators' judgement, could benefit from its use.

DETAILED DESCRIPTION:
The Treatment Use of Domperidone program is also available at the Cleveland Clinic Florida/Weston Gastroenterology Department. This is not a "traditional" research study, but an expanded use protocol for patients who may benefit from the drug. Because of this, this study is enrolling patients via invitation only, and as such, all expenses associated with the drug, initiation and follow up of treatment are the responsibility of the patient or the patient's third party payer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 and older
* Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.
* Patients must have a comprehensive evaluation to eliminate other causes of their symptoms.
* Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

  * increased prolactin levels
  * extrapyramidal side effects
  * breast changes
  * cardiac arrhythmias including QT prolongation and death
  * There is a potential for increased risk of adverse events with the drugs listed in the domperidone protocol addendum.

Exclusion Criteria:

* History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.
* Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc> 450 milliseconds for males, QTc>470 milliseconds for females).
* Clinically significant electrolyte disorders.
* Gastrointestinal hemorrhage or obstruction
* Presence of a prolactinoma (prolactin-releasing pituitary tumor).
* Pregnant or breast feeding female
* Known allergy to domperidone

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio